CLINICAL TRIAL: NCT00913380
Title: Negative Appendectomy Rate Following Low-dose CT vs. Standard-dose CT
Brief Title: Diagnosis of Acute Appendicitis: Low-dose Computed Tomography (CT) Versus Standard-dose CT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: GE Healthcare (Industry); National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Kyoung Ho Lee, Dr., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SNUBH-LDCTinAPPY
Record Dates: First submitted 2009-05-15; First posted 2009-06-04 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-dose CT (Experimental)
  Interventions: Radiation: Diagnostic CT
- Standard-dose CT (Active Comparator)
  Interventions: Radiation: Diagnostic CT

INTERVENTIONS:
Radiation: Diagnostic CT — 2 mSv in an average patient (Low-dose (1/4 to 1/5 of standard-dose))
  Other Names: low-dose CT
  Arms: Low-dose CT
Radiation: Diagnostic CT — 8 mSv in an average patient (Standard-dose CT)
  Other Names: standard-dose CT
  Arms: Standard-dose CT

SUMMARY:
The purpose of this study is to determine whether low-dose CT is not inferior to standard-dose CT in the rate of unnecessary appendectomy.

DETAILED DESCRIPTION:
Acute appendicitis is a very common disease with the lifetime incidence of 7%. Abdomen CT is an established first-line diagnostic test in patients suspected of having acute appendicitis. Since many individuals suspected of having acute appendicitis are young, with a mean age of 30 years, CT radiation is of particular concern.

The estimated lifetime attributable risk of death from cancer due to the radiation exposure of a single abdomen CT study is 2-7/10,000 for average adults ranging 20-40 years in age.

The purpose of this study is to determine whether low-dose CT is not inferior to standard-dose CT in the negative appendectomy rate.

ELIGIBILITY:
Inclusion Criteria:

* Suspected of having acute appendicitis
* Referred for abdomen CT from Emergency Department

Exclusion Criteria:

* Body mass index < 18.5 kg/m2 (ultrasonography is favored)
* Intravenous contrast-enhancement is contraindicated

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 891 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Ho Lee, MD, Principal Investigator — Seoul National University Bundang Hospital; Kyuseok Kim, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim K, Kim YH, Kim SY, Kim S, Lee YJ, Kim KP, Lee HS, Ahn S, Kim T, Hwang SS, Song KJ, Kang SB, Kim DW, Park SH, Lee KH. Low-dose abdominal CT for evaluating suspected appendicitis. N Engl J Med. 2012 Apr 26;366(17):1596-605. doi: 10.1056/NEJMoa1110734. PMID 22533576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: September 2009 to January 2011 Types of location: an emergency department in an urban tertiary hospital in Korea
Pre-assignment Details: None of the enrolled participants were excluded from the trial before assignment to group.
Groups:
- Low-dose CT: Aimed to 2 mSv in an average patient
- Standard-dose CT: Aimed to 8 mSv in an average patient
Period: CT Examination
Arm/Group | Low-dose CT | Standard-dose CT
Started | 444 | 447
Completed | 444 | 447
Not Completed | 0 | 0
Period: Clinical Outcomes
Arm/Group | Low-dose CT | Standard-dose CT
Started | 444 | 447
Completed | 438 | 441
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose CT | Standard-dose CT | Total
Number analyzed (Participants) | 444 | 447 | 891
Age Continuous [Median (Inter-Quartile Range); unit: year]
  Age (year) | 29 [21.5 to 36] | 30 [22 to 37] | 30 [22 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 263 | 539
  Male | 168 | 184 | 352
Race/Ethnicity, Customized [Number; unit: participants]
  Korean | 441 | 445 | 886
  Non-Korean | 3 | 2 | 5
Body mass index [Number; unit: kg/m^2]
  < 18.5 (underweight) | 62 | 60 | 122
  18.5-24.9 (normal) | 312 | 301 | 613
  ≥ 25.0 (overweight to extremely obese) | 70 | 86 | 156
White blood cell [Median (Inter-Quartile Range); unit: x10^3/mm^3] | 10.7 [7.8 to 14.1] | 10.8 [8.0 to 14.3] | 10.8 [7.9 to 14.2]
Segmented neutrophil [Median (Inter-Quartile Range); unit: Percentage of peripheral Leukocytes] | 77.0 [65.8 to 85.2] | 77.3 [65.5 to 83.9] | 77.3 [65.7 to 84.6]
C-reactive protein [Median (Inter-Quartile Range); unit: mg/dL] | 0.5 [0.3 to 2.5] | 0.7 [0.3 to 3.3] | 0.6 [0.3 to 3.1]
CT scanner [Number; unit: participants]
  16-detector CT | 177 | 191 | 368
  64-detector CT | 154 | 144 | 298
  256-detector CT | 113 | 112 | 225
Radiologist [Number; unit: participants]
  Abdominal radiologist | 217 | 225 | 442
  Non-abdominal radiologist | 227 | 222 | 449

OUTCOME MEASURES:

1. Primary Outcome: Negative Appendectomy
Description: Number of participants with unnecessary appendectomies (removal of un-inflamed appendix)
Time Frame: 1 week after surgery
Population: Participants who underwent non-incidental appendectomy. Intention to treat. Complete case analysis.
Measure: Number; unit: participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 172 | 186
participants
  Negative appendectomy | 6 | 6
  Not negative appendectomy | 166 | 180

2. Secondary Outcome: Additional Imaging Test(s)
Description: Number of participants who need additional imaging test(s) to diagnose or rule out appendicitis
Time Frame: 1 week after CT
Population: All participants included in outcome analyses. Intention to treat. Complete case analysis.
Measure: Number; unit: participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 438 | 441
participants
  Additional imaging | 14 | 7
  No additional imaging | 424 | 434

3. Secondary Outcome: Appendiceal Perforation
Description: Number of participants with appendiceal perforation
Time Frame: 1 week after surgery
Population: Participants confirmed to have appendicitis. Intention to treat. Complete case analysis.
Measure: Number; unit: participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 166 | 180
participants
  Perforation | 44 | 42
  No perforation | 122 | 138

4. Secondary Outcome: Interval Between CT and Appendectomy
Description: Time interval between the CT acquisition and non-incidental appendectomy
Time Frame: 1 day after surgery
Population: Participants who underwent non-incidental appendectomy. Intention to treat. Complete case analysis.
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 172 | 186
hr | 7.1 [4.3 to 11.7] | 5.6 [3.4 to 9.2]

5. Secondary Outcome: Interval Between CT and Discharge Without Surgery
Description: Time interval between the CT acquisition and discharge without surgery
Time Frame: 3 months after CT
Population: Participants who did not undergo surgery. Intention to treat. Complete case analysis.
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 249 | 246
hr | 2.5 [1.5 to 4.2] | 2.4 [1.4 to 4.4]

6. Secondary Outcome: Interval From CT to Discharge After Appendectomy
Description: Time interval between the CT acquisition and discharge after appendectomy
Time Frame: 3 months after CT
Population: Participants who underwent non-incidental appendectomy. Intention to treat. Complete case analysis.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 172 | 186
day | 3.4 [2.7 to 4.1] | 3.2 [2.5 to 4.1]

7. Secondary Outcome: Likelihood of Appendicitis in CT Report in Patients Confirmed as Having Appendicitis
Description: Grade 1. Definitely absent. Clinical observation is recommended. Grade 2. Probably absent. Clinical observation is recommended. Grade 3. Indeterminate. Clinical observation or surgical exploration is recommended.
  Grade 4. Probably present. Surgical exploration is recommended. Grade 5. Definitely present. Surgical exploration is recommended. The data is used to calculate sensitivity, specificity, area under receiver-operating-curve and to measure diagnostic confidence.
Time Frame: 3 months after CT
Population: Participants confirmed to have appendicitis. Intention to treat. Complete case analysis.
  There can be missing data if CT report was not made following predefined structured format.
Measure: Number; unit: participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 166 | 180
participants
  Grade 1 | 2 | 4
  Grade 2 | 7 | 5
  Grade 3 | 13 | 11
  Grade 4 | 53 | 34
  Grade 5 | 90 | 126
  Missing | 1 | 0

8. Secondary Outcome: Likelihood of Appendicitis in CT Report in Patients Confirmed as Not Having Appendicitis
Description: Grade 1. Definitely absent. Clinical observation is recommended. Grade 2. Probably absent. Clinical observation is recommended. Grade 3. Indeterminate. Clinical observation or surgical exploration is recommended.
  Grade 4. Probably present. Surgical exploration is recommended. Grade 5. Definitely present. Surgical exploration is recommended. The data are used to calculate sensitivity, specificity, area under receiver-operating-curve and to measure diagnostic confidence.
Time Frame: 3 months after CT
Population: Participants confirmed not to have appendicitis. Intention to treat. Complete case analysis.
  There can be missing data if CT report was not made following predefined structured format.
Measure: Number; unit: participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 272 | 261
participants
  Grade 1 | 185 | 206
  Grade 2 | 65 | 38
  Grade 3 | 11 | 11
  Grade 4 | 3 | 3
  Grade 5 | 4 | 2
  Missing | 4 | 1

9. Other Pre Specified Outcome: Radiation Dose
Description: Radiation dose is measured in terms of dose-length product (mGy•cm) as displayed in the CT console. The "length" indicates the scan range.
Time Frame: 1 day after CT
Population: All participants who underwent CT. Intention to treat. Complete case analysis.
Measure: Median (Inter-Quartile Range); unit: mGy•cm
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 444 | 447
mGy•cm | 116 [94 to 124] | 521 [448 to 564]

10. Other Pre Specified Outcome: Estimate of Carcinogenic Risk Induced by CT Radiation
Description: Age- and sex-specific carcinogenic risk induced by CT radiation. This is not an actual measurement but an estimate of the stochastic risk, based on assumption and calculation from radiation dose used.
Time Frame: 1 day after CT
Reporting Status: Not Posted
Measure: Number; unit: Event per 100,000 persons

11. Secondary Outcome: Diagnosis of Appendiceal Perforation in CT in Patients With Confirmed Appendicitis.
Description: True positive: Perforation was rated as present in CT report and confirmed as present.
  False positive: Perforation was rated as present in CT report and confirmed as absent.
  True negative: Perforation was rated as absent in CT report and confirmed as absent.
  False negative: Perforation was rated as absent in CT report and confirmed as present.
  The data are used to calculate sensitivity and specificity.
Time Frame: 3 months after CT
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 166 | 180
participants
  True positive | 16 | 23
  False positive | 11 | 17
  True negative | 110 | 121
  False negative | 28 | 19
  Missing | 1 | 0

12. Secondary Outcome: Visualization of the Normal Appendix
Description: Grade 0. Not identified Grade 1. Unsure or partly visualized Grade 2. Clearly and entirely visualized
Time Frame: 3 months after CT
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 272 | 261
participants
  Grade 0 | 18 | 13
  Grade 1 | 41 | 20
  Grade 2 | 209 | 227
  Missing | 4 | 1

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Low-dose CT | Standard-dose CT
Serious Adverse Events (participants affected / at risk) | 13/444 | 11/447
Other Adverse Events (participants affected / at risk) | 1/444 | 1/447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose CT (N=444) | Standard-dose CT (N=447)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 6 (6)
Ileus (Gastrointestinal disorders) | 4 (4) | 4 (4)
Wound complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose CT (N=444) | Standard-dose CT (N=447)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
In this diagnostic trial, participants have a variety of abdominal diseases. Events with CTCAE v4 Grade 2 or less are not considered reportable according to the Study Protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes